CLINICAL TRIAL: NCT05721079
Title: Prophylactic Use of Extracorporeal Photopheresis (ECP) After Lung Transplantation
Brief Title: Extracorporeal Photopheresis (ECP) After Lung Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Peter Jaksch, Priv.Doz. Dr., Priv.-Doz.Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECP-LUTX V 3.0
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Lung Transplant Infection; Lung Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ECP with standard triple IS (Experimental)
  Interventions: Device: ECP (Extracorporeal Photopheresis System)
- standard triple IS (Active Comparator)
  Interventions: Device: ECP (Extracorporeal Photopheresis System)

INTERVENTIONS:
Device: ECP (Extracorporeal Photopheresis System) — Patients who are assigned to the ECP group receive treatments by means of the THERAKOS ® CELLEX ® Photopheresis System (Mallinckrodt Pharmaceuticals Inc.) with either double- or single-needle access. During the leukapheretic processing, 1500 ml of whole blood is processed, and peripheral blood mononuclear cells (MCNs) are separated by centrifugation and collected in the buffy coat. 8-methoxypsoralen (Uvadex®, Mallinckrodt Pharmaceuticals Inc.) at a dose of 20 μg/ml is added to the MNC collection bag and cells are irradiated with ultraviolet A light (1.5 J/cm2) in a 1-mm-thick film through a photoactivation plate. After exposure of the cells to the ultraviolet light, the buffy coat is reinfused into the patient.
  Other Names: 8-Methoxypsoralen

SUMMARY:
The purpose of this study is to investigate the use of ECP for lung-transplanted patients to reduce the occurrence of acute and chronic rejection and CMV-infection.

DETAILED DESCRIPTION:
The intention of the planned study is the use of ECP as a form of induction treatment in combination with standard triple-drug immunosuppressive therapy (IS). This is a single-center prospective randomized controlled trial conducted at Medical University of Vienna between 2018 and 2020. It includes 31 COPD recipients per group. Treatment group underwent ECP with in addition to IS after lung transplantation. Control group received only IS. The primary outcome was a composite outcome defined as incidence of high-grade ACR, CMV infection or CLAD within 24 months after lung transplantation.

Parallel to the clinical parameters, immunologic investigations will be performed to get a better insight into the mechanisms of ECP on the immune system. The dynamics of Tregs and dentritic cell will be analyzed to compare the influence of ECP vs standard IS.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first lung transplantation
* Patient underlying disease COPD
* Male or female be 18 years or older
* Patients (male and female) must agree to use an acceptable method of birth control the treatment period of 3 months and 3 months afterward
* Patients must have a body weight more than 40 kg
* Patients must have a platelet count more than 20.000/cmm
* Patients must be willing and capable of understanding the purpose and risks of the study and must sign a statement of informed consent

Exclusion Criteria:

* Previous organ transplantation
* Women who are pregnant and/or lactating
* Patients with hypersensitivity or allergy to both heparin and citrate products
* Patients who are unable to tolerate extracorporeal volume shifts associated with ECP treatment due to the presence of any of the following conditions: uncompensated congestive heart failure, pulmonary edema, renal failure or hepatic failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Composite endpoint | 24 months
  the incidence of high-grade ACR, cytomegalovirus (CMV) infection or CLAD

SECONDARY OUTCOMES:
Frequency of ACR and of lymphocytic bronchiolitis (LB) | 24 months
  Frequency of ACR and of lymphocytic bronchiolitis (LB)
Incidence of clinically treated infections | 24 months
  Incidence of clinically treated infections
Detection of plasma CMV DNA | 24 months
  Detection of plasma CMV DNA
Patient survival | 36 months
  Patient survival
Graft survival | 36 months
  Graft survival
Incidence of de-novo donor specific antibodies | 24 months
  Incidence of de-novo donor specific antibodies
Number of AMR episodes | 24 months
  Number of AMR episodes
Incidence of CLAD | 36 months
  Incidence of CLAD

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
To evaluate the safety and efficacy of ECP in addition to a standard triple immunosuppressive therapy consisting of Tacrolimus (Tac), Mycophenolate Mofetile (MMF) and corticosteroids to prevent rejection and infections.
Supporting Information: Study Protocol, SAP
Time Frame: Available for the next 6 months